CLINICAL TRIAL: NCT03692897
Title: An Observational Study of Patients With Chronic Hepatitis B (CHB) Infection
Status: Terminated | Type: Observational
Why Stopped: Study Closure
Sponsor: Target PharmaSolutions, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TARGET-HBV
Record Dates: First submitted 2018-09-04; First posted 2018-10-02 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Hepatitis B; Hepatitis; Liver Diseases
MeSH Terms: conditions — Hepatitis B; Hepatitis; Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Patients enrolled in TARGET-HBV may be invited to participate in the Biorepository Bank (BSB). Blood samples for biomarker and DNA assays will be collected on a voluntary basis and participation in this project will not affect participation in the main study. These samples will be shipped to a central repository for storage to use in future studies. Samples stored at the biorepository will be identified only with the participant's unique study ID number and the date the sample was obtained. The link between the participant's study ID number and their name will be available only at the site where the samples were obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: All approved therapies for the treatment of Chronic Hepatitis B (CHB) — All approved therapies for the treatment of Chronic Hepatitis B (CHB).

SUMMARY:
The TARGET-HBV study engages an observational research design to conduct a comprehensive review of outcomes for patients with CHB infection. The initial phase of the study that enrolled patients treated with tenofovir alafenamide (TAF) was successfully completed. The current protocol (Amendment 1) describes the second phase of the study that will engage research activities for patients being managed for CHB in usual clinical practice in the US and Canada. The study addresses important clinical questions regarding the management of CHB by collecting and analyzing data from patients at academic and community medical centers. TARGET-HBV creates a robust database of real-world data regarding the natural history, management, and health outcomes related to antiviral treatments used in clinical practice.

ELIGIBILITY:
Inclusion

1. Male or female patients, age ≥18 years
2. Being managed for chronic hepatitis B (CHB), including patients who have achieved functional cure and patients with concurrent delta hepatitis

Exclusion

1. Inability to provide written informed consent
2. Known history of Human Immunodeficiency Virus (HIV)
3. History of liver transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 5,000 adult Chronic Hepatitis B (CHB) patients in the US and Canada; the first 500 patients enrolled were patients in the US with a medical history of tenofovir alafenamide (TAF) use for the treatment of chronic HBV.
Sampling Method: Non-Probability Sample
Enrollment: 1708 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
Natural history of CHB: Characteristics of CHB infection | Up to 10 years
Natural history of CHB: Participant demographics | Up to 10 years
Natural history of CHB: Treatment use | Up to 10 years
Natural history of CHB: Treatment response | Up to 10 years
Time point of clinical response | Every 6 months for 10 years
Natural history of CHB: Disease progression | Up to 10 years
Adverse event frequency and severity | Up to 10 years

SECONDARY OUTCOMES:
Reasons for treatment discontinuation | Up to 10 years

CONTACTS AND LOCATIONS:
Locations (31):
- United States (30):
  - Banner University Medical Center Phoenix, Phoenix, Arizona
  - Asian Pacific Liver Center at Coalition of Inclusive Medicine, Los Angeles, California
  - California Liver Research Institute, Pasadena, California
  - Stanford University, Redwood City, California
  - UC Davis GI/Hepatology Clinical Trials Unit, Sacramento, California
  - Silicon Valley Research Institute, San Jose, California
  - Yale University Digestive Diseases, New Haven, Connecticut
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - University of Miami, Schiff Center for Liver Disease, Miami, Florida
  - Consultative Gastroenterology, Atlanta, Georgia
  - Atlanta Gastroenterology, Atlanta, Georgia
  - Rush Universtiy Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Mercy Medical Center, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Minnesota Gastroenterology, P.A., Plymouth, Minnesota
  - Rutgers, Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Dreamwork Medical, PLLC, Flushing, New York
  - Northwell Health Center for Liver Diseases and Transplantation, Manhasset, New York
  - NYU Langone Health, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Columbia University Medical Center, New York, New York
  - UNC Liver Center, Chapel Hill, North Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - Digestive and Liver Disease Specialist, Norfolk, Virginia
  - Bon Secours Liver Institute of Richmond, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Swedish Organ Transplant and Liver Center, Seattle, Washington
  - University of Washington/Harborview Medical Center, Seattle, Washington
- UHN Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bernstein DE, Trinh HN, Schiff ER, Smith CI, Mospan AR, Zink RC, Fried MW, Lok AS. Safety and Effectiveness of Tenofovir Alafenamide in Usual Clinical Practice Confirms Results of Clinical Trials: TARGET-HBV. Dig Dis Sci. 2022 Jun;67(6):2637-2645. doi: 10.1007/s10620-021-07033-y. Epub 2021 May 31. PMID 34059991